CLINICAL TRIAL: NCT01819025
Title: Face-to-face CBT Treatment of Depression With Smartphone Support
Brief Title: Cognitive Behavioral Therapy Treatment of Depression With Smartphone Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-PC-HH-KHL
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: Depression; Behavioral activation; Smartphone application; Face-to-face; Blended therapy
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 face-to-face and smartphone-app (Experimental): Four face-to-face therapy sessions and smartphone app as a complement and support to the four sessions.
  Interventions: Behavioral: 4 face-to-face therapy session and a smartphone-app
- TAU (Active Comparator): 10 sessions of face-to-face therapy, full behavioral activation
  Interventions: Behavioral: CBT, treatment as usual

INTERVENTIONS:
Behavioral: 4 face-to-face therapy session and a smartphone-app — An 8 week blended therapy with both face-to-face therapy sessions and support through a smartphone application.
  Arms: 4 face-to-face and smartphone-app
Behavioral: CBT, treatment as usual — 10 sessions of face-to-face therapy, full behavioral activation
  Arms: TAU

SUMMARY:
The purpose of this study is to investigate whether face-to-face Cognitive Behavioral Therapy (CBT) with a smartphone application, focused on providing support in homework assignments and an increase in behavioral activation, is effective in treating mild to moderate depression. The study will be conducted as a randomized controlled treatment study investigating the effect of the current blended treatment compared to treatment as usual.

DETAILED DESCRIPTION:
Mild to moderate depression is a major health problem, which lowers the quality of life for the individual and generates enormous costs for society. Several forms of psychotherapy have been found to be effective in the treatment of depression. Among these, behavioral activation has a strong empirical base. The efficacy of behavioral activation for treating major depressive disorders has been established in a number of studies over the last four decades.

Moreover face-to-face treatments could benefit from using smartphones as an adjunct to the regular sessions, which in the case of behavioral activation treatments for depression could facilitate activity scheduling and homework, which are crucial elements of the treatment. It may also be possible to reduce the number of sessions.

Since it has been shown that full behavioral activation is an effective treatment for mild to moderate depression, this study will be designed as a so-called non-inferiority study in which the treatment group, given fewer meetings face-to-face, but instead support in the form of a smartphone application. Instead of a traditional behavioral activation treatment of 10 sessions, the treatment group will be given four face-to-face CBT sessions and a smartphone app as a complement and support to the four sessions. As a control, the investigators will give full behavioral activation with 10 sessions of face-to-face therapy.

ELIGIBILITY:
Inclusion Criteria:

* depressive symptoms according to DSM-IV
* have access to a smartphone and to the Internet
* have good knowledge of the Swedish language

Exclusion Criteria:

* recent (during last 6 weeks) change in psychiatric medication
* presently in any other psychological treatment
* severe depression
* suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Beck Depression Inventory (BDI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.

SECONDARY OUTCOMES:
Quality of Life Inventory (QOLI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Acceptance & Action Questionnaire (AAQ)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Beck Anxiety Inventory (BAI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P)- Change from baseline | Two weeks pre treatment and at six months post treatment.
  Change from baseline in health cost burden and at six months post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Ly KH, Topooco N, Cederlund H, Wallin A, Bergstrom J, Molander O, Carlbring P, Andersson G. Smartphone-Supported versus Full Behavioural Activation for Depression: A Randomised Controlled Trial. PLoS One. 2015 May 26;10(5):e0126559. doi: 10.1371/journal.pone.0126559. eCollection 2015. PMID 26010890